CLINICAL TRIAL: NCT02003066
Title: Effect of Goal-directed Fluid Therapy Using Stroke Volume Variation in Patients Undergoing Free Flap Reconstruction After Head and Neck Cancer Resection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4-2013-0638
Record Dates: First submitted 2013-11-18; First posted 2013-12-06 (Estimated); Last update posted 2019-01-28 (Actual); Status verified 2019-01

CONDITIONS: General Anesthesia
Keywords: Fluid Therapy; Head and Neck Neoplasms; Surgical Flaps
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard (Experimental)
  Interventions: Procedure: Standard fluid therapy
- Conservative (Active Comparator)
  Interventions: Procedure: Conservative fluid therapy

INTERVENTIONS:
Procedure: Standard fluid therapy — In Standard fluid therapy group, the administration of fluid will be guided to maintain mean blood pressure more than 65 mmHg, urine output more than 0.5 ml/kg/hr, and central venous pressure less than 14 mmHg.
  Arms: Standard
Procedure: Conservative fluid therapy — In Goal directed fluid therapy group, the administration of fluid will be guided by stroke volume variation. The anesthesiologist will infuse volulyte (Fresenius Kabi, Bad Homburg, Germany) 200 ml if stroke volume variation is over 12%. If cardiac index is below 2.5 l/min/m2 and stroke volume variation is below 12%, start dobutamine.
  Arms: Conservative

SUMMARY:
Investigators hypothesized that goal-directed fluid therapy using stroke volume variation will improve postoperative recovery in patients undergoing free flap reconstruction after head and neck cancer resection. Investigators will compare the effect of goal-directed fluid therapy using stroke volume variation on recovery in patients undergoing free flap reconstruction after head and neck cancer resection.

ELIGIBILITY:
Inclusion Criteria:

* adult patients of age over 20 years scheduled for free flap reconstruction after head and neck cancer resection

Exclusion Criteria:

* valvular heart disease
* congestive heart failure
* liver failure
* renal failure
* pregnant woman
* allergy to hydroxyethyl starch solutions
* coagulation abnormalities

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2014-03-20 (Actual); Primary Completion 2016-03-08 (Actual); Study Completion 2016-03-08 (Actual)

PRIMARY OUTCOMES:
Length of hospital stay | 1 month after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Yonsei University Health System, Seoul, South Korea

REFERENCES:
- [Derived] Kim HJ, Kim EJ, Lee HJ, Min JY, Kim TW, Choi EC, Kim WS, Koo BN. Effect of goal-directed haemodynamic therapy in free flap reconstruction for head and neck cancer. Acta Anaesthesiol Scand. 2018 Aug;62(7):903-914. doi: 10.1111/aas.13100. Epub 2018 Mar 25. PMID 29574681